CLINICAL TRIAL: NCT01249352
Title: A Phase II, Randomized, Controlled, Open-Label Study Comparing Standard Chemoradiation Versus Chemoradiation Associated with Nimotuzumab As the Treatment of Locally Advanced Esophageal Cancer
Brief Title: A Study of Chemoradiation Associated with Nimotuzumab As the Treatment of Locally Advanced Esophageal Cancer
Acronym: NICE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF024-201
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2025-03-31 (Actual); Status verified 2014-01

CONDITIONS: Esophageal Cancer; Adenocarcinoma
Keywords: Esophageal Cancer; Nimotuzumab; EF024; EF024-201
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma | interventions — nimotuzumab; Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STANDARD CHEMORADIATION (Active Comparator): Cisplatin 75 mg/m2, IV IV doses on D1 of each chemotherapy cycle, for 4 cycles Fluorouracil 1000 mg/m2, IV IV doses in a 24-hour continuous infusion, from D1 to D4 of each chemotherapy cycle, for 4 cycles.
  Radiotherapy 50.4 Gy, fractions of 1.8 Gy/day Equivalent to 28 fractions for 5 and a half weeks.
  Interventions: Drug: Nimotuzumab; Drug: Cisplatin; Drug: Fluorouracil; Radiation: Radiotherapy
- CHEMORADIATION + NIMOTUZUMAB (Experimental): Nimotuzumab 200 mg, IV weekly IV doses for up to 26 weeks. Cisplatin 75 mg/m2, IV IV dose on D1 of each chemotherapy cycle, for 4 cycles, always after nimotuzumab.
  Fluorouracil 1000 mg/m2, IV IV dose in a 24-hour continuous infusion, from D1 to D4 of each chemotherapy cycle, for 4 cycles.
  Radiotherapy 50.4 Gy, fractions of 1.8 Gy/day Equivalent to 28 fractions for 5 and a half weeks.
  Interventions: Drug: Nimotuzumab; Drug: Cisplatin; Drug: Fluorouracil; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Nimotuzumab — 200 mg, IV Weekly IV dose for up to 26 weeks.
Drug: Cisplatin — 75 mg/m2, IV dose on D1 of each chemotherapy cycle, for 4 cycles, always after nimotuzumab.
Drug: Fluorouracil — 1,000 mg/m2, IV dose in a 24-hour continuous infusion, from D1 to D4, every chemotherapy cycle, for 4 cycles.
Radiation: Radiotherapy — Radiotherapy 50.4 Gy, fractions of 1.8 Gy/day

SUMMARY:
The primary objective of this study is to assess the efficacy of nimotuzumab in combination with chemotherapy and radiotherapy for the treatment of locally advanced esophageal cancer, comparing it to that of the conventional treatment with radiation and chemotherapy.

The secondary objective of this study is to assess the health-related quality of life for the nimotuzumab in combination with chemotherapy and radiotherapy regimen, compared to the standard chemoradiation regimen in the treatment of inoperable locally advanced esophageal cancer.

DETAILED DESCRIPTION:
This will be a phase II, randomized, controlled, open-label, multicenter, and two-arm study. The study will be conducted in Brazil and has the purpose of determining the activity and safety of nimotuzumab in terms of overall survival, TTP, clinical and endoscopic response rates, resectability rate, toxicity profile, and quality of life. All participating patients will sign a consent form before they undergo any study-related procedure. The eligible patients will have locally advanced esophageal cancer, and they will be randomized to one of two treatment groups. Randomization will be centrally coordinated by the sponsor and performed by means of the electronic CRF itself.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Histological prove of SCC or esophageal adenocarcinoma;
3. T1N1M0, T2N1M0, T3N0M0, T4N0M0, T3N1M0, T4N1M0, qqTqqNM1a stage, according to the TNM system42;
4. Life expectation above 6 months;
5. Inoperable superior, medial, or distal third esophageal cancer, including GE junction tumors, defined as type I and II tumors in the Siewert classification43 (see Appendix B);
6. Performance status 0, 1, or 2, according to the Eastern Cooperative Oncology Group criteria44 (ECOG) (see Appendix C);
7. Creatinine clearance ≥ 60 ml/min, according to the Cockcroft and Gault formula45 (see Appendix D);
8. Adequate body functions, indicated by

   * Creatinine clearance ≥ 60 ml/min;
   * Bilirubin, transaminase, alkaline phosphatase, and gamma-GT < 1,5 x the upper limit of normal;
   * leucocytes ≥ 3000/μl;
   * granulocytes ≥ 1500/ μl;
   * hemoglobin ≥ 9 g/dl;
   * platelets ≥ 80000/ μl;
9. Adequate calorie ingestion, at the investigator's discretion;
10. He/she must have signed the informed consent form

Exclusion Criteria:

1. Previous or planned treatment of esophageal carcinoma with surgery, radiotherapy, chemotherapy, or antineoplastic biological therapy;
2. Presence of active infection;
3. Knowledge of the presence of HIV seropositivity;
4. Presence of severe comorbidities that, in the investigator's opinion, will put the patient at a significantly higher risk or will damage the protocol compliance;
5. Presence of a significant neurological or psychiatric disease, including dementia and seizures, as per the investigator's judgment;
6. History of malignant neoplasm, except for adequately treated skin basal carcinoma or SCC, and cervical carcinoma in situ;
7. Presence of peripheral neuropathy;
8. Knowledge of the presence of hypersensitivity or allergy to drugs that will be administered in this protocol;
9. History of severe allergic reaction;
10. Pregnancy or lactation;
11. Presence of aerodigestive fistula (trachea and/or bronchia);
12. Evident presence of trachea and/or bronchia infiltration by the tumor;
13. Presence of uncontrolled hypercalcaemia ≥ 2.9 mmol/L (or grade >1, according to the NCI-CTCAE, version 3.0).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Overall survival and assessment of the complete endoscopic response | 2 years
  The primary endpoint of this study is the overall survival at the end of Phase II. At the end of Phase II, the assessment of the complete endoscopic response, and the regimen safety will be used to decide if the study will continue to Phase III.

SECONDARY OUTCOMES:
Complete clinical response rate | 2 years
  * Time to tumor progression (TTP);
  * Complete clinical response rate, defined as the proportion of patients with absence of visible disease in the high endoscopy and in the chest and abdomen computerized tomography, in the population assessable for response;
  * Complete endoscopic response rate, defined as the absence of visible disease in the high endoscopy;
  * Resectability rate;
  * Safety:
  * Quality of life, according to the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire;
  * Relationship between efficacy and safety and the tumor characteristics.

CONTACTS AND LOCATIONS:
Locations (19):
- Brazil (19):
  - Hospital Evangélico do Cachoeiro do Itapemirim, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital Universitário de Brasília, Brasília, Federal District
  - Santa Casa de Misericórdia de BH, Belo Horizonte, Minas Gerais
  - Hospital Erasto Gaetner, Curitiba, Paraná
  - Hospital Geral de Bonsucesso, Rio de Janeiro, Rio de Janeiro
  - Instituto Nacional do Câncer (INCA), Rio de Janeiro, Rio de Janeiro
  - Hospital da cidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - Centro de Novos Tratamentos de Itajaí, Itajaí, Santa Catarina
  - Hospital Municipal São José, Joinville, Santa Catarina
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Centro Oncológico Mogi das Cruzes, Mogi das Cruzes, São Paulo
  - Faculdade de Medicina do ABC / CEPHO, Santo André, São Paulo
  - Centro de Estudos de Investigações Clíncas (CEIC), São Caetano do Sul, São Paulo
  - Hospital de Base, São José do Rio Preto, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
  - Hospital São Paulo (UNIFESP), São Paulo, São Paulo
  - Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo

REFERENCES:
- [Derived] de Castro Junior G, Segalla JG, de Azevedo SJ, Andrade CJ, Grabarz D, de Araujo Lima Franca B, Del Giglio A, Lazaretti NS, Alvares MN, Pedrini JL, Kussumoto C, de Matos Neto JN, Forones NM, Fernandes Junior HJ, Borges G, Girotto G, da Silva IDCG, Maluf-Filho F, Skare NG. A randomised phase II study of chemoradiotherapy with or without nimotuzumab in locally advanced oesophageal cancer: NICE trial. Eur J Cancer. 2018 Jan;88:21-30. doi: 10.1016/j.ejca.2017.10.005. Epub 2017 Nov 24. PMID 29179134